CLINICAL TRIAL: NCT02820584
Title: A Phase I Study of Immunotherapy With GSC -Loaded Dendritic Cells in Patients With Recurrent Glioblastoma
Acronym: DENDR-STEM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DENDR-STEM
Record Dates: First submitted 2016-02-22; First posted 2016-07-01 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: de Novo Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSC-loaded autologous dendritic cells (Experimental): DC-GSC immunotherapy. Six vaccinations are envisaged. The first three vaccinations will be performed every two weeks; subsequent three vaccinations every month. The first vaccination will be performed using 20 million DC, the second and third with 10 million DC; and from the 4th vaccine 5 million DC
  Interventions: Biological: GSC-loaded autologous dendritic cells

INTERVENTIONS:
Biological: GSC-loaded autologous dendritic cells

SUMMARY:
Mono-center, un-controlled, open label, first in human, clinical trial. Approximately 20 patients (in order to achieve 12 valuable patients). The expected accrual time would range between 12 and 18 months. Follow-up, including clinical, immune and radiological monitoring will end two years after the initial surgery of the last patient enrolled. The primary objective will be to assess the activity of immunotherapy in terms of its effect on immune response. In particular we will investigate the effect of treatment on effector cells including CD8 T cells, NK cells and Natural Killer T (NKT) cells. The sample size of 12 eligible patients was identified on ethical and practical considerations, rather than by a formal sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years;
* Histological diagnosis of de novo GBM (i.e. not secondary GBM);
* Gross total resection as evaluated by MRI performed within 72 hours from surgery;
* Karnofsky Performance Status (KPS) ≥60 at the time of first progression;
* Written informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding;
* Participation in other clinical trials with experimental drugs simultaneously;
* Mandatory treatment with corticosteroids or salicylates in anti-inflammatory dose;
* Presence of sub-ependymal diffusion of the tumor;
* Presence of multi-focal GBM lesion;
* Haematology: leukocytes (WBC) < 3x103/μl, absolute lymphocyte count< 0.5x103/μl, Absolute neutrophil count (ANC) < 1x103/μl, hemoglobin< 9 g/dL, platelets< 50x103/μl within two days prior to leukapheresis;
* AST (SGOT)/ALT (SGPT) ≥3 X institutional Upper Limit Normal (ULN) at the time of leukapheresis;
* Serum creatinine>1.5 ULN or calculated creatinine clearance < 60 ml/min at time of surgery;
* Documented immune deficiency;
* Documented systemic autoimmune disease;
* Positivity for HBV, HIV, HCV, Treponema Pallidum;
* Allergies to any component of the DC vaccine;
* Other active malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety: - incidence, nature, severity and seriousness of AEs, according to NCI-CTCAE version 4.0; - maximum toxicity grade and percentage of patients experiencing grade 3-4 by each patient for each specific toxicity; - patients with at least a SAE. | 18 months
  Safety will be assessed as follows:
  * Incidence, nature, severity and seriousness of AEs, according to NCI-CTCAE, version 4.0
  * Maximum toxicity grade experienced by each patient for each specific toxicity
  * Percentage of patients experiencing grade 3-4 toxicity for each specific toxicity
  * Patients with at least a SAE
  * Patients with at least a SADR
  * Patients with at least a Suspected Unexpected Serious Associated Reaction (SUSAR).
Incidence, severity and type of AEs throughout the study, and toxicities will be graded according to the National Cancer Institute Common Toxicity Criteria for AE (CTCAE), version 4.0 | 18 months

SECONDARY OUTCOMES:
Probability to obtain the full vaccine dosage, i.e. the percentage of patients who will be treated with at least 2 vaccine injections. | 18 months
Immunologic activity | 18 months
  activity of immunotherapy in terms of its effect on immune response of predefined immune effector cells.
Progression free survival (PFS) | 18 months
  Progression Free Survival after immunotherapy is defined for each patient as the time of onset of immunotherapy to the date of second progression.
Quality of life | 18 months
  Treatment effect on quality of life will be assessed using the EORTC QLQ-C30 and BN-20.
Quality of life | 18 months
  Treatment effect on quality of life will be assessed using the BN-20 questionnaire.
Overall survival (OS) | 18 months
  Overall Survival after immunotherapy is defined for each patient as the time of onset of immunotherapy to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Finocchiaro, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico "Carlo Besta" di Milano

IPD SHARING:
Plan to Share IPD: No